CLINICAL TRIAL: NCT05415943
Title: An Open-label, Multicentre, Single-arm Safety and Efficacy Clinical Investigation of Diagnostic Microprobe (inPROBE) for the Assessment of HER2 Receptor Expression in Population of Women at High Risk of Breast Cancer
Brief Title: Safety and Efficacy Assessment of Diagnostic Microprobe (inPROBE) in Women at High Risk of Breast Cancer (Part I Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SDS Optic S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SDS-HER-01-2018
Record Dates: First submitted 2022-06-07; First posted 2022-06-13 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women at high risk of breast cancer (Experimental): Women with a confirmed diagnosis of breast cancer by thick-needle biopsy and known HER2 receptor expression status, referred for surgical treatment.
  Interventions: Device: Diagnostic microprobe (inPROBE) medical device

INTERVENTIONS:
Device: Diagnostic microprobe (inPROBE) medical device — Introduction of the inPROBE microprobe (two simultaneous punctures) into the breast as a procedure prior to surgical resection of tumors with known HER2 receptor status.

SUMMARY:
The purpose of this study is to preliminarily determine the correlation of HER2 receptor levels detected with the inPROBE diagnostic probe relative to receptor status as determined by standard methods (IHC/FISH), in women with both HER2-positive and HER2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent to participate in the clinical investigation;
2. Female patient aged ≥ 18 to ≤ 75 years;
3. The patient's overall health status as determined by Eastern Cooperative Oncology Group (ECOG) from 0 to 1;
4. Preserved full ability to communicate with the investigator and to understand and comply with the requirements of the Clinical investigation plan;
5. High likelihood of attending follow-up appointments in accordance with the study design and completing this study in accordance with this Clinical investigation plan.
6. The presence of a malignant neoplasm (breast cancer) confirmed by histopathologic examination of material from a gross needle biopsy of the tumor, with specific HER2 receptor status.
7. Patient referred for surgical treatment of breast cancer.

Exclusion Criteria:

1. History of treatment with trastuzumab, or other HER 2 receptor-binding antibody, as part of neoadjuvant (induction) therapy for currently diagnosed and treated breast cancer.
2. A skin disorder that prevents or contraindicates to perform a probe examination in the opinion of the investigator;
3. Breast inflammation/infection on the day of the probe examination;
4. Allergy to any component of the medical device that is the subject of this clinical investigation;
5. An implant in the breast where the inPROBE study and surgery will be performed;
6. Any physical or psychiatric condition, or laboratory test values outside the normal range, which in the opinion of the investigator constitute a contraindication to the patient's participation in this clinical investigation or pose a risk of exclusion from the study or premature termination of participation in the study;
7. Any clinically significant abnormality in physical examination, vital signs, or laboratory tests that, in the opinion of the investigator, is a contraindication to participation in this clinical trial;
8. Pregnancy or breastfeeding;
9. Participation in another clinical trial within 30 days prior to signing informed consent to participate in this clinical investigation;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Preliminary determination of HER2 receptor concentration ranges detected with inPROBE corresponding to HER2 receptor status (positive/negative) as determined by current diagnostic standard (IHC/FISH). | Day 1

SECONDARY OUTCOMES:
The occurrence of defects, failures, and fractures of the inPROBE probe during the diagnostic procedure leading to AE/ SAE. | Day 1 - Day 14
Comparison of the correlation of HER2 receptor concentrations detected by the inPROBE probe located in the tumor and in the immediate tumor area in HER2 positive patients. | Day 1

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Uniwersyteckie Centrum Leczenia Chorób Piersi, Szpital Uniwersytecki w Krakowie, Krakow
  - Klinika Chirurgii Onkologicznej, Lublin